CLINICAL TRIAL: NCT03076021
Title: Effects of Isotretinoin on CYP2D6 Activity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Mary Hebert, Professor of Pharmacy, Adjunct Professor of Obstetrics and Gynecology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00002324; R01GM124264 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: CYP2D6 Polymorphism
MeSH Terms: interventions — Isotretinoin; Dextromethorphan

STUDY DESIGN:
Intervention Model Description: Prospective, pre-post drug interaction study evaluating an approved drug (Phase 4) with a Phase 1 study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adolescents (Other): dextromethorphan pre- and post isotretinoin
  Interventions: Drug: Isotretinoin; Drug: dextromethorphan

INTERVENTIONS:
Drug: Isotretinoin — Drug interaction study
  Other Names: accutane
Drug: dextromethorphan — Drug interaction study
  Other Names: robitussin pediatric

SUMMARY:
Specific Aim: To investigate if isotretinoin (13-cis-retinoic acid) administration decreases CYP2D6 activity in adolescent patients.

DETAILED DESCRIPTION:
In this aim, we will conduct a drug-drug interaction study evaluating the effects of 13-cis-retinoic acid on non-induced CYP2D6 activity in adolescent patients. Secondary analysis will evaluate the relationship between retinoid concentrations and CYP2D6 activity in these special populations

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant
* ≥ 12 years
* Patients with severe acne that are expected to receive isotretinoin for therapeutic reasons

Exclusion Criteria:

* Weight < 80 lbs
* Allergy or adverse reaction to dextromethorphan, vitamin A or isotretinoin
* Pregnant or planning to become pregnant
* Unable to follow isotretinoin risk evaluation and mitigation strategies (REMS) program (also known as iPLEDGE program)
* Chronic or persistent cough accompanying asthma, smoking or chronic obstructive pulmonary disease,
* Productive cough,
* Fever,
* Known kidney disease,
* Known liver disease,
* Diabetes
* Obesity, body mass index ≥ 30 kg/m2
* Bipolar disease,
* Attention deficit disorder,
* Social phobia,
* Concurrent or use within 14 days of drugs known to interact with dextromethorphan or cytochrome P450 2D6 (CYP2D6) or drugs known to increase the risk of adverse effects from dextromethorphan
* Concurrent use of any other product containing dextromethorphan
* Consuming foods, beverages or dietary supplements known to interact with dextromethorphan or CYP2D6
* Unable to give written informed consent/assent,
* Inability to fast for 4 hours prior to study.
* Wards of the State

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Hebert, PharmD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, we plan to follow NIGMS/NIH and University of Washington requirements for data sharing.

REFERENCES:
- [Result] Zhao Y, Vary JC Jr, Yadav AS, Czuba LC, Shum S, LaFrance J, Huang W, Isoherranen N, Hebert MF. Effect of isotretinoin on CYP2D6 and CYP3A activity in patients with severe acne. Br J Clin Pharmacol. 2024 Mar;90(3):759-768. doi: 10.1111/bcp.15938. Epub 2023 Nov 21. PMID 37864393

RESULTS

PARTICIPANT FLOW:
Groups:
- Individuals Expected to Receive Isotretinoin for Therapeutic Reasons: Each subject had 2 study days, one pre-isotretinoin treatment and one while receiving isotretinoin.
Period: Pre-isotretinoin
Arm/Group | Individuals Expected to Receive Isotretinoin for Therapeutic Reasons
Started | 33
Completed | 33
Not Completed | 0
Period: Isotretinoin
Arm/Group | Individuals Expected to Receive Isotretinoin for Therapeutic Reasons
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects that completed the study.
Groups:
- Study Group: Individuals expected to receive isotretinoin for therapeutic reasons
Arm/Group | Study Group
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — Collected directly from subjects
  years | 23.5 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: CYP2D6 Activity as Measured by the Molar Concentration Ratio of Dextromethorphan (DM)/Dextrophan (DX)
Description: dextromethorphan (DM)/dextrophan (DX) molar concentration Metabolic Ratio. The metabolic ratio is unit-less as the molar concentrations cancel out.
Time Frame: 1 week to 6 months
Population: The number of subjects included in the analysis is less than the number that completed the study because only cytochrome P450 extensive metabolizers were included in the analysis. Each person served as their own control (pre-isotretinoin and with isotretinoin). Pre-isotretinoin study was completed prior to starting isotretinoin and then the same study was completed after the subject had been on isotretinoin for 1 week to 6 months.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Pre-isotretinoin: Individuals expected to receive isotretinoin for therapeutic reasons
- With Isotretinoin: Individuals receiving isotretinoin for therapeutic reasons.
Arm/Group | Pre-isotretinoin | With Isotretinoin
Number analyzed (Participants) | 24 | 24
Ratio | 16.0 [10.2 to 25.0] | 12.5 [8.9 to 17.6]

ADVERSE EVENTS:
Time Frame: 1 week to 6 months
Arm/Group | Pre-isotretinoin | With Isotretinoin
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03076021/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03076021/SAP_001.pdf
  • Informed Consent Form (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03076021/ICF_002.pdf